CLINICAL TRIAL: NCT05379114
Title: Comparative, Monocentric Study for the Evaluation of the Non-inferiority of a New Medical Device on the Treatment of Head Lice Infestation
Brief Title: Comparative Study for the Evaluation of a New Medical Device on the Treatment of Head Lice Infestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Perrigo CSCI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20E4084
Record Dates: First submitted 2022-05-06; First posted 2022-05-18 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Head Lice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INVESTIGATIONAL DEVICE (Experimental): new medical device for the treatment of head lice infestation: Paranix ®
  Interventions: Other: INVESTIGATIONAL DEVICE
- COMPARATOR DEVICE (Active Comparator): dimethicone based head lice treatment (medical device class 1) already in market in europe: Pouxit ®
  Interventions: Other: Comparator device

INTERVENTIONS:
Other: INVESTIGATIONAL DEVICE — new medical device for the treatment of head lice infestation: Paranix ®
  Arms: INVESTIGATIONAL DEVICE
Other: Comparator device — well established medical device for the treatment of head lice infestation (dimethicone based) - Pouxit ®
  Arms: COMPARATOR DEVICE

SUMMARY:
Pediculosis capitis or head lice infestation is a human medical condition caused by the infestation of the hair by the parasitic insect Pediculus humanus capitis (human head lice). The most common symptom of infestation is pruritus (itching) on the head which normally intensifies 3 to 4 weeks after the initial infestation.

The test item has been developed with the ambition to offer a complete head lice treatment, whilst also offering ultimate convenience in use - making treatment of head lice infestation easy, and effective in few minutes.

The objectives of this clinical study are to assess the efficacy and the safety of a new Medical Device for lice infestation treatment compared to a comparator device, already in market.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject;
2. Sex: male or female;
3. Age: 2 years and above;
4. Subject with a slight to moderate lice infestation
5. Subjects with various hair type (from 1 to 3C - hair scale) and hair length (from short to mid length hair, not exceeding shoulder)
6. Documented oral informed consent for all subjects, including minors, given freely and expressly before the start of the study
7. Written informed consent for subjects ≥18 years or legal guardian for subjects< 18 years given freely and expressly before start of the study;
8. Written assent for subjects ≥12 to <18 years.
9. Subject/Subject's legal guardian is psychologically able to understand the study related information and to give written informed consent;
10. Females of childbearing potential must have a negative pregnancy test before the beginning of the study

Exclusion Criteria:

In terms of population

1. Pregnant (confirmed by pregnancy test for women of childbearing potential) or nursing woman or planning a pregnancy during the study;
2. Subject who had been deprived of their freedom by administrative or legal decision or adult subject who is under guardianship;
3. Subject in a social or sanitary establishment;
4. Subject in an exclusion period from a previous study or who is currently participating to another study on hair/scalp or who participated to another clinical study on hair/scalp within 3 months before first visit.
5. Subject suspected to be non-compliant according to the Investigator's judgment.
6. Subject with curly or frizzy hair (type 4a to 4c in the hair type scale above)
7. Subject with hair length below the shoulder.
8. Subjects with more than 24 lice on the head

   In terms of associated pathology
9. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
10. Subject with a cutaneous disease on the studied zone (scalp and hair).
11. Subject with severe scratches or open wounds/skin damages on the scalp (lice bites allowed however).
12. Subject with a known or suspected allergy to any of the components/materials of the investigational or comparator devices, anti-lice comb or post-treatment shampoo.
13. Subject who has diabetes (type 1 or 2).
14. Subject with known or suspected immune deficiency or autoimmune disease.

    Relating to previous or ongoing treatment
15. Subject undergoing a topical treatment on the test area or a systemic treatment with :

    * anti-inflammatory medication and/or anti-histamines during the previous 2 weeks and during the study;
    * corticosteroids during the 2 previous weeks and during the study;
    * retinoids and/or immunosuppressors during the 3 previous months and during the study;
    * any medication stabilized for less than one month.
16. Subject who received an anti-lice treatment in the previous 2 months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Cure Rate after complete treatment | day 7
  The cure rate is defined as the rate of subjects having no live lice on scalp 7 days after the last application of the product.
Cure Rate after complete treatment | day 14
  The cure rate is defined as the rate of subjects having no live lice on scalp 7 days after the last application of the product.

SECONDARY OUTCOMES:
Cure rate after one dose of Investigational device (ID) | Day 7
  Comparison of the percentage of subjects cured after one dose of the investigational device compared to the percentage of subjects cured with two doses of the comparator device.
Dead and live lice/nymphs and number of eggs after combing | Day 0 and Day 7 if applicable
  Number of dead and live lice/nymphs and number of eggs collected on the anti-lice comb after treatment
Live lice and nymphs, after application | Day 1 and Day 8 if applicable
  Evaluation of the presence of live lice and nymphs, for both groups, without combing on scalp
Number of participants with treatment-related adverse events as assessed by investigator | Day 0, 7, 8 and 14 if applicable
  Evaluation of the safety and tolerability of the investigational device versus comparator
Subject reported perceived acceptability, effectiveness and subjective evaluation assessed via questionnaire data | Day 7 or Day14
  Evaluation of the perceived acceptability, effectiveness and subjective evaluation.
  Subject perception questionnaire with the following scale items:
  totally agree agree rather agree rather disagree disagree

CONTACTS AND LOCATIONS:
Locations (1):
- Céline Lhéritier, Quatre Bornes, Mauritius

IPD SHARING:
Plan to Share IPD: No